CLINICAL TRIAL: NCT06017596
Title: Evaluation of Polyetheretherketone (PEEK) Framework Inserted in Multiunit Abutments of All-on-4 Concept for the Mandibular Edentulous Arch.
Brief Title: CAD-CAM PEEK Framework for All-on-4 Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A17100221
Record Dates: First submitted 2023-08-05; First posted 2023-08-30 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-07

CONDITIONS: Bone Loss
Keywords: All-on-Four implant; CAD-CAM; PEEK framework
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PEEK group (Experimental): Patients received PEEK framework prosthesis
  Interventions: Device: PEEK framework

INTERVENTIONS:
Device: PEEK framework — All-on-4 implants with PEEK framework of fixed detachable prosthesis

SUMMARY:
This study was conducted to evaluate the clinical peri-implant soft tissue changes during the first year after occlusal loading and the ridge base relation after 3 years for mandibular computer-aided design and computer-aided manufacturing (CAD/CAM) screw-retained implant-supported hybrid prosthesis of polyetheretherketone (PEEK) framework utilized with All-on-Four treatment concept.

DETAILED DESCRIPTION:
Sixteen completely edentulous patients were rehabilitated by four implants following the All-on-Four protocol. After 3 months, the definitive prosthesis was constructed to be a screw-retained CAD-CAM milled framework from the modified PEEK (BioHPP), bonded to polymethylmethacrylate teeth and a pink-shaded indirect light-polymerized nano-filled composite resin imitating the soft tissues. Peri-implant soft tissue changes regarding plaque, bleeding, gingival scores, and probing depth were evaluated at prosthesis insertion (T0), 6 months (T1), and 12 months (T2) after insertion. Also, monitoring of the ridge base relation was performed using cone-beam computed tomography CBCT at the time of insertion (T0), and 1 year (T1), 2 years (T2), and 3 years (T3) after mandibular fixed detachable All-on-Four framework insertion.

ELIGIBILITY:
Inclusion Criteria:

* Completely edentulous maxillary and mandibular ridges with sufficient mandibular bone height in the inter-foraminal area confirmed with panoramic x-rays.
* All selected patients will be with sufficient inter-arch space and restorative space.
* All selected patients will have apparently healthy ridge covered by compressible oral mucosa and free from any ridge flabbiness.

Exclusion Criteria:

* Patients with systemic diseases that contraindicate implant placement such as hematologic diseases, serious problems of coagulation and diseases of the immune system. Also, metabolic diseases related to bone resorption such as uncontrolled diabetics or osteoporosis will be also excluded
* History of para-functional habits (Bruxism, clenching), smoking and alcoholism.
* History of radiation therapy in the head and neck region.

Ages: 60 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2023-02-12 (Actual); Study Completion 2023-03-20 (Actual)

PRIMARY OUTCOMES:
evaluation of changes in the peri-implant soft tissue health | six months
  Peri-implant soft tissue changes regarding plaque scores were assessed using the modified plaque index
evaluation of changes in the peri-implant soft tissue health | six months
  Peri-implant soft tissue changes regarding bleeding scores were assessed using the bleeding index.
evaluation of changes in the peri-implant soft tissue health | six months
  Peri-implant soft tissue changes regarding the gingival scores were assessed using the simplified gingival index.

SECONDARY OUTCOMES:
Ridge base relation monitoring | 3 years
  periodic monitoring of the changes in the alveolar ridge height in millimeters using CBCT

CONTACTS AND LOCATIONS:
Overall Officials: Khloud Ezzat, PhD, Principal Investigator — Lecturer of Prosthodontics
Locations (1):
- Khloud Ezzat, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No